CLINICAL TRIAL: NCT05661175
Title: A Comparative Study of One-handed Lithotripsy and Traditional Lithotripsy in Percutaneous Nephrolithotomy
Brief Title: Application of One-handed Lithotripsy in Percutaneous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of University of South China (Other)
Responsible Party: Principal Investigator, Li Mingyong, MD, Associate professor, The First Affiliated Hospital of University of South China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USCKF202011K20
Record Dates: First submitted 2022-12-02; First posted 2022-12-22 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Percutaneous Nephrolithotomy
Keywords: Percutaneous nephrolithotomy; one-handed lithotripsy; Urinary calculi; traditional PCNL
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to an experimental or control group in parallel.
Who Masked: Participant
Masking Description: A single-blind trial in which participants were unaware of the study group and the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group(group 1) (Experimental): Percutaneous nephrolithotripsy was performed using one - hand lithotripsy
  Interventions: Procedure: one-handed technique
- Control group(group 2) (No Intervention): Percutaneous nephrolithotripsy was performed using traditional techniques

INTERVENTIONS:
Procedure: one-handed technique — Traditional percutaneous nephrolithotripsy usually requires the left hand to hold the nephroscope and the right hand to control the fiber for lithotripsy.Our intervention is to control the depth and direction of the sheath with the left hand, the nephroscope in the right hand and control the fiber optic lithotripsy
  Arms: Experimental group(group 1)

SUMMARY:
Percutaneous nephrolithotomy(PCNL) is a surgical method for upper urinary calculi.Traditional percutaneous nephrolithotomy usually requires the lithotripsy with the left hand holding the nephroscope and the right hand adjusting the laser fiber,which requires a lot of practice to master this technique.The goal of this study is to explore the safety and effectiveness of the PCNL with one-handed lithotripsy technique

DETAILED DESCRIPTION:
This is a key clinical research project of the University of South China(NO.USCKF201902K01).The goal of this study is to compare the safety,effectiveness and feasibility between the percutaneous nephrolithotomy with one-handed technique and the traditional percutaneous nephrolithotomy in the treatment of upper urinary calculi. It is a prospective, randomized controlled single center study that is conducted for 2 years anticipatively. The clinic physician is responsible for patient recruitment and allocation.For random allocation,participants are randomly grouped by coin toss method.Participants with front side are assigned to experimental group,where they undergo PCNL with one-handed lithotripsy.Participants with reverse side are assigned to control group and undergo traditional PCNL.The doctors managing the operations accept participants and execute the surgical treatments.All participants sign clinical-trial informed consent and surgical informed consent during the preoperative conversation.Follow-up observation is conducted for 1 month after surgery. After completion of the study, we collect relevant clinical data from the participants. The primary and secondary outcomes are analyzed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants who met the the applications of PCNL surgery in the 2019 Chinese Guidelines for the Diagnosis and Treatment of Urological Disease.
* Participants who agree to undergo one-hand lithotripsy.

Exclusion Criteria:

* Obvious surgical contraindications, such as severe heart and lung insufficiency, abnormal coagulatory function.
* Confirmation by computerized tomography (CT) images and blood biochemical indicators of infectious stones or complex staghorn stones

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-11-03 (Estimated); Study Completion 2023-11-03 (Estimated)

PRIMARY OUTCOMES:
Operative time | during the procedure
  From the completion of anesthesia to the end of the suture incision.
Stone clearance rate | Day 2 after the surgery
  Preoperative and postoperative stone dimensions are compared by radiological assessment. Postoperative residual calculi < 4 mm in diameter reflect complete removal of calculi (stone-free rate = 100%)
Renal pelvis mucosal injury rate | during the procedure
  Number of accidental injuries of renal pelvis mucosa during operation
Changes in renal bleeding after surgery | Hour 3 after the surgery
  Pre- vs. post-operative difference in hemoglobin and hematocrit values

SECONDARY OUTCOMES:
Hospital costs | immediately after the discharge
  The cost from hospitalization to discharge.
Hospital stay | immediately after the discharge
  The number of days from hospitalization to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mingyong Li, MD, Principal Investigator — The First Affiliated Hospital of University of South China
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 1 year after publication.
Access Criteria: When proper editing or review requirements are met, the study data will be available from the study manager after the study is completed.

DOCUMENTS (1):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT05661175/Prot_000.pdf